CLINICAL TRIAL: NCT01500421
Title: The Øresund Copenhagen-Malmø Acute Stroke Cooling Trial
Brief Title: Safty and Feasibility Study of Therapeutic Cooling in Acute Ischemic Stroke (COOLAID Øresund)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Malmö University (Other)
Responsible Party: Principal Investigator, Derk W. Krieger MD, Ph.D, Principal Investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-D-2008-105
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2011-12-28 (Estimated); Status verified 2011-12

CONDITIONS: Cerebral Infarction
Keywords: Hypothermia, Induced
MeSH Terms: conditions — Cerebral Infarction; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- TH - Endovacular alone (Experimental): Patients randomized to this arm are cooled to a bodytemperature of 33 degrees with an endovascular groin catheter (Copenhagen only).
  Interventions: Device: TH - Endovascular alone (Alsius®, Zoll, USA)
- TH - Endovascular + nasopharyngeal induction (Experimental): Patients randomized to this arm are cooled to a bodytemperature of 33 degrees with endovascular catheter along with nasopharyngeal induction (Copenhagen only).
  Interventions: Device: TH - Endovascular + nasopharyngeal induction (Alsius®, Zoll, USA) (Rhinochill®, Benechill, USA)
- Standard Treatment (No Intervention): Patients are treated with standard care in the stroke ward.
- TH - Surface Cooling (Experimental): Patients randomized to this arm are cooled to a bodytemperature of 33 degrees with cold saline infusion followed by surface cooling with Arctic Sun Cooling system, Medivance, USA (Malmø only)
  Interventions: Device: Intravenous cold saline and surface cooling (Arctic Sun, Medivance, USA)

INTERVENTIONS:
Device: TH - Endovascular alone (Alsius®, Zoll, USA) — Patients are cooled with an endovascular (Alsius®, Zoll, USA) groin catether (9,3 french).
  Arms: TH - Endovacular alone
Device: TH - Endovascular + nasopharyngeal induction (Alsius®, Zoll, USA) (Rhinochill®, Benechill, USA) — Patient are cooled with a groin endovascular catheter (Alsius®, Zoll, USA) + a nasopharyngeal induction catheter (Rhinochill®, Benechill, USA) in the nostrils. The nasopharyngeal induction is designed to give a more quick and localised brain cooling.
  Arms: TH - Endovascular + nasopharyngeal induction
Device: Intravenous cold saline and surface cooling (Arctic Sun, Medivance, USA) — Infusion of ice cold saline of 4°C (25 mL/kg body weight)followed by surface cooling
  Other Names: Arctic Sun, Medivance, USA
  Arms: TH - Surface Cooling

SUMMARY:
This study is designed to investigate the safty and feasibility of therapeutic hypothermia in acute stroke patients. Soon after arrival in the stroke unit patients are randomized to either hypothermia in the intensive care unit (ICU) or standard treatment in the stroke ward.

Patients randomized to therapeutic hypothermia are analgo-sedated and cooled to at temperature of 33 degrees for a period of 24 hours.

DETAILED DESCRIPTION:
Ischemic stroke remains a diagnosis with limited treatment opportunities and a treatment with the ability to target patients outside the normal treatment window is wanted.

Therapeutic hypothermia (TH) treatment has long been recognised as a treatment of patients with global ischemia following caridac arrest.

This trial is designed to address the safty and feasibility of TH in acute stroke patients.

Patients arriving in our stroke ward are observed for 3 hours. Only non-remitting patients are allowed into the trial.

Patients are randomized to either therapeutic hypothermia with endovascular catheter + nasopharyngeal induction or endovascular catheter alone in the intensive care unit (ICU) (in Copenhagen, Denmark) or intravenous cold saline infusion followed by surface cooling (in Malmø, Sweden)versus standard treatment in a stoke unit.

Patients brought to the ICU are sedated and mechanically ventilated.

Therapeutic hypothermia is induced with a endovascular catether and a nasopharyngeal catheter. Body temperature is lowered to 33 degrees and sustained for a period of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* National Institute of Health Stroke Scale (NIHSS) score on admission between 5 and 18
* Inclusion within 24 hours after stroke onset
* Diagnosis of ischemic stroke verified by MRI, CT or CTP adjudicated by including physician
* Informed consent from patient or proxy

Exclusion Criteria:

* Modified ranking scale (mRS)>2 indicating significant disability before onset of stroke
* MRI or CT evidence for massive ischemic damage (>50% Middle cerebral artery (MCA) territory)
* Severe concomitant diseases such as heart failure, chronic obstructive lung disease or known cancer
* Presently on anticoagulation treatment
* No informed consent from patient or proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety | 3 month
  Feasibility and safety defined as mortality and morbidity 3 months after ictus

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 3 months
  mRS score after 7 days and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Background] De Georgia MA, Krieger DW, Abou-Chebl A, Devlin TG, Jauss M, Davis SM, Koroshetz WJ, Rordorf G, Warach S. Cooling for Acute Ischemic Brain Damage (COOL AID): a feasibility trial of endovascular cooling. Neurology. 2004 Jul 27;63(2):312-7. doi: 10.1212/01.wnl.0000129840.66938.75. PMID 15277626
- [Background] Hamann GF, Burggraf D, Martens HK, Liebetrau M, Jager G, Wunderlich N, DeGeorgia M, Krieger DW. Mild to moderate hypothermia prevents microvascular basal lamina antigen loss in experimental focal cerebral ischemia. Stroke. 2004 Mar;35(3):764-9. doi: 10.1161/01.STR.0000116866.60794.21. Epub 2004 Feb 19. PMID 14976330
- [Background] Krieger DW, De Georgia MA, Abou-Chebl A, Andrefsky JC, Sila CA, Katzan IL, Mayberg MR, Furlan AJ. Cooling for acute ischemic brain damage (cool aid): an open pilot study of induced hypothermia in acute ischemic stroke. Stroke. 2001 Aug;32(8):1847-54. doi: 10.1161/01.str.32.8.1847. PMID 11486115
- [Background] Lyden PD, Allgren RL, Ng K, Akins P, Meyer B, Al-Sanani F, Lutsep H, Dobak J, Matsubara BS, Zivin J. Intravascular Cooling in the Treatment of Stroke (ICTuS): early clinical experience. J Stroke Cerebrovasc Dis. 2005 May-Jun;14(3):107-14. doi: 10.1016/j.jstrokecerebrovasdis.2005.01.001. PMID 17904009
- [Background] Milhaud D, Thouvenot E, Heroum C, Escuret E. Prolonged moderate hypothermia in massive hemispheric infarction: clinical experience. J Neurosurg Anesthesiol. 2005 Jan;17(1):49-53. PMID 15632543
- [Background] Schwab S, Georgiadis D, Berrouschot J, Schellinger PD, Graffagnino C, Mayer SA. Feasibility and safety of moderate hypothermia after massive hemispheric infarction. Stroke. 2001 Sep;32(9):2033-5. doi: 10.1161/hs0901.095394. PMID 11546893